CLINICAL TRIAL: NCT02995356
Title: Evaluation of the Axonemal Dynein Heavy Chain 5 and Creatine Kinase Concentration in Cervical Fluid for Early Detection of the Ectopic Pregnancy
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Cagdas Sahin, MD, Ege University
Other Study IDs: 2.101.2015.0076
Record Dates: First submitted 2016-12-12; First posted 2016-12-16 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Ectopic Pregnancy
Keywords: Ectopic pregnancy; Axonemal Dynein Heavy Chain 5; Creatine Kinase; Cervical fluid
MeSH Terms: conditions — Pregnancy, Ectopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Doubt for ectopic pregnancy group: This group participants have doubt for ectopic pregnancy in terms of beta-HCG pregnancy follow-up results and ultrasonography results.
  Interventions: Other: Collecting cervical liquid and sera samples
- Normal intrauterine pregnancy group: This groups participants have normal intrauterine pregnancy
  Interventions: Other: Collecting cervical liquid and sera samples

INTERVENTIONS:
Other: Collecting cervical liquid and sera samples

SUMMARY:
Patients who have doubt for ectopic pregnancy will be enrolled for our study. These patients will be determined with using irregular increased human chorionic gonadotropin (beta-HCG) results and no embryo reported ultrasonography results. Plasma and cervical fluid samples will be taken from these patients and axonemal dynein heavy chain 5 and creatine kinase levels of samples will be compared between patients who have doubt for ectopic pregnancy and patients who have intrauterine pregnancy. Concentration of these proteins in samples will be evaluated. If any difference will be found between groups in favour of ectopic pregnancy, these results might be interpreted as these proteins useful for early detecting of the ectopic pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Doubted ectopic pregnancy
* Without any finding about intrauterine pregnancy in ultrasonography results
* Without any vaginal bleeding
* Having irregular pregnancy test results
* Beta-HCG results should be at least upper than 100 milli-International unit (mIU/ml)
* Having fist trimester pregnancy for intrauterine pregnancy group
* Without any emergency findings

Exclusion Criteria:

* Doubted incomplete abortion
* Having vaginal bleeding
* Having ultrasound results which include intrauterine embryo report
* Having lower than 100 mIU/ml beta-HCG results
* Without fetal heart rate in intrauterine pregnancy group
* Having older than fist trimester pregnancy for intrauterine pregnancy group
* Having emergency findings

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who have doubt for ectopic pregnancy will be selected for study group and patients who have intrauterine pregnancy will be selected for control group.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Concentration of Axonemal Dynein Heavy Chain 5 | 1 year
Concentration of creatine kinase | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Medicine Faculty, Department of Obstetrics and Gynecology, Izmir, Turkey (Türkiye)

REFERENCES:
- [Derived] Sahin C, Uygun ZO, Hortu I, Akdemir A, Kocamanoglu M, Ergenoglu AM, Akcay Y. Using dynein heavy chain 5 and creatine kinase levels in cervical fluid and blood for early diagnosing of ectopic pregnancy. J Obstet Gynaecol Res. 2021 Mar;47(3):921-927. doi: 10.1111/jog.14616. Epub 2020 Dec 17. PMID 33336538